CLINICAL TRIAL: NCT07218380
Title: FORAGER-2: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Vepugratinib Combined With Enfortumab Vedotin and Pembrolizumab in Adults With Untreated Locally Advanced or Metastatic Urothelial Carcinoma With an FGFR3 Genetic Alteration
Brief Title: A Study of Vepugratinib (LY3866288) in Participants With Cancer in the Urinary Tract
Acronym: FORAGER-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27333; J4G-MC-JZVD (Other: Eli Lilly and Company); 2025-522855-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-09; First posted 2025-10-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Neoplasm Metastasis
Keywords: FGFR3; Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: There will be an open-label safety lead in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vepugratinib + EV + Pembrolizumab (Safety Lead In) (Experimental): Vepugratinib administered orally with EV + pembrolizumab administered IV
  Interventions: Drug: Vepugratinib; Drug: EV; Drug: Pembrolizumab
- Vepugratinib + Enfortumab Vedotin (EV) + Pembrolizumab (Experimental): Vepugratinib administered orally, and EV + pembrolizumab administered by intravenous (IV) infusion.
  Interventions: Drug: Vepugratinib; Drug: EV; Drug: Pembrolizumab
- Placebo + EV + Pembrolizumab (Placebo Comparator): Placebo administered orally, and EV + pembrolizumab administered by IV infusion.
  Interventions: Other: Placebo; Drug: EV; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Vepugratinib — Administered orally
  Arms: Vepugratinib + EV + Pembrolizumab (Safety Lead In); Vepugratinib + Enfortumab Vedotin (EV) + Pembrolizumab
Other: Placebo — Administered orally
  Arms: Placebo + EV + Pembrolizumab
Drug: EV — Administered by IV infusion
Drug: Pembrolizumab — Administered by IV infusion

SUMMARY:
The purpose of this study is to test a new medicine, vepugratinib, in comparison with placebo, to see if it is safe and can help people with a bladder cancer that is advanced or has spread.

Vepugratinib or placebo will be administered in combination with enfortumab vedotin and pembrolizumab.

Study participation could last up to approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed, unresectable locally advanced or metastatic urothelial cancer (mUC). Individuals with mixed histology other than small cell or neuroendocrine carcinoma are eligible if a urothelial component is present.
* Have a qualifying fibroblast growth factor receptor 3 (FGFR3) genetic alteration determined via molecular testing from a tumor or blood sample obtained at or any time after diagnosis of advanced or metastatic urothelial cancer.
* Have measurable disease by investigator assessment defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Have adequate laboratory parameters

Exclusion Criteria:

* Have received prior systemic therapy for locally advanced or metastatic urothelial cancer (mUC).
* Have any unresolved toxicities greater than Grade 1 Common Terminology Criteria for Adverse Events ([CTCAE] version 5.0) from prior neoadjuvant or adjuvant systemic therapy.
* Have ongoing sensory or motor neuropathy of Grade 2 or higher
* Have untreated or uncontrolled central nervous system (CNS) involvement or any history of leptomeningeal disease.
* Current evidence corneal keratopathy or retinal disorder confirmed by ocular examination at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events related to vepugratinib in combination with EV and pembrolizumab | From baseline up to 90 months
Safety Lead-in: Overall Response Rate (ORR) | From baseline up to 90 months
  ORR by Investigator Assessment.
Progression-free Survival (PFS) | Baseline to Study Completion (estimated as 6 years)
  PFS by blinded independent committee review (BICR).

SECONDARY OUTCOMES:
Safety Lead-in: Disease Control Rate (DCR) | From baseline up to the end of Cycle 2 (each Cycle is 21 days)
  DCR by investigator assessment.
Safety Lead-in: Time to Response (TTR) | From baseline up to 90 months
  TTR by investigator assessment.
Overall Survival (OS) | Baseline to Study Completion (estimated as 6 years)
Objective Response Rate (ORR) by BICR | Baseline to Study Completion (estimated as 6 years)
Duration of Response (DoR) | Baseline to Study Completion (estimated as 6 years)
  DOR by BICR.
Progression-free Survival (PFS) | Baseline to Study Completion (estimated as 6 years)
  PFS by investigator assessment.
Objective Response Rate (ORR) | Baseline to Study Completion (estimated as 6 years)
  Percentage of Participants who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR)ORR by investigator assessment
Duration of Response (DOR) | Baseline to Study Completion (estimated as 6 years)
  DOR by investigator assessment.
Progression-free Survival 2 (PFS2) | Baseline to Study Completion (estimated as 6 years)
  PFS2 by investigator assessment.
Plasma Concentrations of Vepugratinib | Cycle 1 Day 1 to Study completion (estimated as 90 months)
  PK samples are to be drawn every odd cycle while participant on study.
Change from Baseline in Global Health Status/Quality of Life (QOL) and Physical Function Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline to Study Completion (estimated as 6 years)
  The EORTC QLQ-C30 is a validated self-reported general cancer questionnaire consisting of 30 items with a recall of the past 7 days. Response options range from 1) "very poor" to 7) "excellent." Higher scores represent better overall HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (276):
- United States (51):
  - Clearview Cancer Institute, Huntsville, Alabama
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - TRIO-US (Translational Research in Oncology-US), Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Hunt Cancer Institute, an Affiliate of Cedars-Sinai Cancer (TMPN), Torrance, California
  - AdventHealth Medical Group - Porter, Denver, Colorado
  - Colorado West Healthcare System - Grand Valley Oncology, Grand Junction, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - St. Luke's Cancer Institute: Boise, Boise, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Parkview Research Center at Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer -T, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute- Research, Sioux Falls, South Dakota
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - USO-Texas Oncology-Central/South Texas, Austin, Texas
  - World Research Link, Baytown, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Nova Oncology, McAllen, Texas
  - US Oncology Research Network, The Woodlands, Texas
  - USO - Texas Oncology - Northeast Texas, Tyler, Texas
  - USO - Virginia Oncology Associates, Norfolk, Virginia
- Australia (9):
  - Box Hill Hospital, Box Hill
  - Mater Misericordiae Limited, Brisbane
  - GenesisCare - Campbelltown, Campbelltown
  - Austin Health, Heidelberg
  - Macquarie University, Macquarie University
  - Sir Charles Gairdner Hospital, Perth
  - Prince of Wales Hospital, Randwick
  - Western Health-Sunshine & Footscray Hospitals, St Albans
  - Calvary Mater Newcastle, Waratah
- Brazil (25):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - CPAM - Centro de Pesquisas da Amazônia, Belém
  - Oncocentro de Minas Gerais, Belo Horizonte
  - Hospital Mario Penna, Belo Horizonte
  - Hospital Tacchini, Bento Gonçalves
  - Centro Integrado de Oncologia de Curitiba, Curitiba
  - IOP Pesquisa, Curitiba
  - Centro Paraibano De Oncologia - Oncoclínicas, João Pessoa
  - Hospital de Cancer de Londrina, Londrina
  - Liga Norte Riograndense Contra o Câncer, Natal
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Clinica Amo - Rio Vermelho, Salvador
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul
  - Centro de Oncologia - CEON+ - Unidade São Caetano do Sul, São Caetano do Sul
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital BP, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Centro Paulista de Oncologia Clínica, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary
  - Hamilton Health Sciences-Juravinski Cancer Centre, Hamilton
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus, Québec
  - BC Cancer Vancouver, Vancouver
- China (25):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Cancer hospital, Beijing
  - Beijing GoBroad Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Chongqing University Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Sun Yat-Sen University Cancer Centre, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Ningbo First Hospital, Ningbo
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
- Czechia (6):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Fakultni nemocnice Motol, Prague
- Denmark (5):
  - Aalborg Universitetshospital, Syd, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen
  - Næstved Sygehus, Næstved
- France (12):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU de Bordeaux Hop St ANDRE, Bordeaux
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHRU de Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon Cedex08
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nîmes - Institut de Cancérologie du Gard - Hôpital Universitaire Carém -T, Nîmes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Oncopole Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (25):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Evangelisches Krankenhaus Bielefeld - Johannesstift, Bielefeld
  - Johanniter-Krankenhaus, Bonn
  - Studienzentrum Bayenthal Urologische Partnerschaft Köln, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden
  - Urologicum Duisburg Fachärztesozietät - Walsum, Duisburg
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - NCT, Heidelberg
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Rechts Der Isar Der Technischen Universität München, Munich
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Studienpraxis Urologie, Nürtingen
  - Universitätsmedizin Rostock, Rostock
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Italy (8):
  - Instituto Tumori Giovanni Paolo II, Bari
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Istituto Nazionale Tumori Regina Elena, Rome
- Japan (20):
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Hirosaki University Hospital, Hirosaki
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - St. Marianna University Hospital, Kawasaki
  - Kagawa University Hospital, Kita-ku
  - Kobe City Medical Center General Hospital, Kobe
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Gunma Prefectural Cancer Center, Otashi
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho
  - Tokushima University Hospital, Tokushima
  - Tsukuba University Hospital, Tsukuba
- Netherlands (4):
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (12):
  - IN VIVO, Bydgoszcz
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie, Koszalin
  - Pratia MCM Krakow, Krakow
  - AIDPORT Sp. z o.o., Skórzewo
  - GYNCENTRUM Szpital, Sosnowiec
  - Luxmed Onkologia sp. z o. o., Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw
  - WSD MEDI, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Szpital Grochowski im. dr med. Rafała Masztaka SPZOZ, Warsaw
  - Wojskowy Instytut Medyczny Państwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wrocaw
- South Korea (10):
  - National Cancer Center, Goyang-si
  - Chungnam national university hospital, Junggu
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (26):
  - Hospital Infanta Cristina, Badajoz
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Institut Català d'Oncologia (ICO) - Girona, Girona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario Marqués de Valdecilla, Santander
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Arnau de Vilanova, Valencia
- Taiwan (11):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center (NTUCC), Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (11):
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Sakarya University School of Medicine, Adapazarı
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Dr. Lutfi Kirdar Kartal Training and Research Hospital, Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul
  - zmir Katip Çelebi Üniversitesi Atatürk Eitim Ve Aratrma Hastanesi, Izmir
- United Kingdom (7):
  - Huddersfield Royal Infirmary, Huddersfield
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Royal Marsden Hospital (Sutton), London
  - Royal Marsden Hospital (Chelsea), London
  - The Christie NHS Foundation Trust, Manchester
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Trials site — https://trials.lilly.com/en-US/trial/661564